CLINICAL TRIAL: NCT02173249
Title: A Single-Center, Open-Label, Study of the Plasma Pharmacokinetics and Safety of AC-170 0.24%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aciex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-100-0007
Record Dates: First submitted 2014-06-13; First posted 2014-06-24 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Healthy

ARMS (1):
- AC 170 0.24% (Experimental)
  Interventions: Drug: AC 170 0.24%

INTERVENTIONS:
Drug: AC 170 0.24% — 1 drop in each eye 2 times daily for 1 week

SUMMARY:
The purpose of this study is to evaluate the Plasma Pharmacokinetics and Safety of AC 170 0.24% in Healthy, Adult Subjects when used twice daily for one week.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 and no older than 55 years of age
* be able to self-administer eye drops or have a parent/legal guardian available for this purpose
* have blood and urine analysis within normal limits
* have ocular health within normal limits

Exclusion Criteria:

* known contraindications or sensitivities to the study medication or its components
* have any active systemic or ocular disorder (other than refractive disorder)
* have inability to comply with controlled diet
* have used prescription or non prescription drugs within washout period and throughout study
* have used alcohol or tobacco within the washout period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cmax values of AC 170 0.24% | 1 week
  Plasma samples will be drawn at specified time points and then analyzed to determine Cmax values of AC 170 0.24% in the plasma
Tmax values of AC 170 0.24% | 1 week
  Plasma samples will be drawn at specified time points and then analyzed to determine Tmax values of AC 170 0.24% in the plasma
AUC values of AC 170 0324% | 1 week
  Plasma samples will be drawn at specified time points and then analyzed to determine AUC values of AC 170 0.24% in the plasma
T 1/2 values of AC 170 0.24% | 1 week
  Plasma samples will be drawn at specified time points and then analyzed to determine T 1/2 values of AC 170 0.24% in the plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States